CLINICAL TRIAL: NCT00416624
Title: RC05CB A Pilot, Randomized Comparison of Standard Weekly Epoetin Alfa to Every-3-Week-Epoetin Alfa and Every 3-Week Darbepoetin Alfa
Brief Title: Epoetin Alfa or Darbepoetin Alfa in Treating Patients With Anemia Caused by Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000522677; P30CA015083 (NIH); RC05CB (Other: Mayo Clinic Cancer Center & MCCRC); 06-002991 (Other: Mayo Clinic IRB); EPOANE3015 (Other: Centocor protocol)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2015-09

CONDITIONS: Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; extramedullary plasmacytoma; isolated plasmacytoma of bone; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; Waldenstrom macroglobulinemia; post-transplant lymphoproliferative disorder; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; anemia; monoclonal gammopathy of undetermined significance; primary systemic amyloidosis; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; mast cell leukemia; adult nasal type extranodal NK/T-cell lymphoma; untreated hairy cell leukemia
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Waldenstrom Macroglobulinemia; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Lymphoma, Extranodal NK-T-Cell | interventions — Darbepoetin alfa; Epoetin Alfa; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Epoetin alfa - 40000 units (Experimental): 40,000 Units
  Interventions: Drug: darbepoetin alfa; Drug: epoetin alfa; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment
- Epoetin alfa - 80000 units (Experimental): 80,000 Units
  Interventions: Drug: darbepoetin alfa; Drug: epoetin alfa; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment
- Epoetin alfa - 120000 Units (Experimental): 120,000 Units
  Interventions: Drug: darbepoetin alfa; Drug: epoetin alfa; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment
- Darbepoetin alfa*** (Experimental): 500 mcg
  Interventions: Drug: darbepoetin alfa; Drug: epoetin alfa; Procedure: fatigue assessment and management; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: darbepoetin alfa
Drug: epoetin alfa
Procedure: fatigue assessment and management
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Epoetin alfa and darbepoetin alfa may cause the body to make more red blood cells. They are used to treat anemia caused by chemotherapy in patients with cancer.

PURPOSE: This randomized clinical trial is studying four different schedules of epoetin alfa or darbepoetin alfa to compare how well they work in treating patients with anemia caused by chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the relative efficacy of four different erythropoietic agent dosing schedules comprising epoetin alfa or darbepoetin alfa, in terms of the proportion of patients with chemotherapy-associated anemia who achieve a weekly and overall hematopoietic response.

Secondary

* Compare the effect of these regimens on the mean hemoglobin increment measured weekly from baseline to 15 weeks in patients with a baseline hemoglobin of less than or equal to 10.5 g/dL.
* Compare the time required to achieve hemoglobin levels within the goal range 11.0-12.0 g/dL in patients treated with these regimens.
* Compare the effect of these regimens on the proportion of patients requiring red blood cell transfusions and on the number of transfusions required.
* Compare the weekly change in hemoglobin in patients treated with these regimens.
* Compare the need for dose reduction in patients treated with these regimens.
* Compare the adverse event profiles of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, unblinded, pilot study. Patients are stratified according to severity of anemia (mild [hemoglobin ≥ 9.5 g/dL] vs severe [hemoglobin < 9.5 g/dL]), platinum-containing regimen (yes vs no), and tumor type (nonmyeloid hematologic malignancy vs solid tumor). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive epoetin alfa subcutaneously (SC) on day 1. Treatment repeats weekly for up to 15 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive epoetin alfa SC on day 1 (at a higher dose than in arm I). Treatment repeats every 3 weeks for up to 5 courses in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive epoetin alfa SC on day 1 (at a higher dose than in arm II). Treatment repeats every 3 weeks for up to 5 courses in the absence of disease progression or unacceptable toxicity.
* Arm IV: Patients receive darbepoetin alfa SC on day 1. Treatment repeats every 3 weeks for up to 5 courses in the absence of disease progression or unacceptable toxicity.

Hemoglobin levels are monitored throughout the study on a weekly basis and before each drug dose is administered. Drug dosing is adjusted (e.g., held, reduced, resumed at a lower dose) as needed to maintain hemoglobin values within the desired ranges.

Quality of life is assessed at baseline and at weeks 4, 7, 10, 13, and 16.

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 320 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor or nonmyeloid hematologic malignancy (e.g., plasma cell dyscrasia or lymphoproliferative disorder)

  * No nonmelanomatous skin cancer
* Hemoglobin ≤ 10.5 g/dL
* Ferritin > 20 ng/mL (i.e., not obviously iron deficient)
* Planning to receive ≥ 12 weeks of anticancer chemotherapy

  * Biological therapy (e.g., hypomethylating agents, monoclonal antibodies, or small molecule pathway inhibitors) with an individual or cumulative regimen incidence of grade 3 or 4 anemia > 10% is considered chemotherapy for purposes of this study
* No known anemia secondary to any of the following:

  * Cyanocobalamin (vitamin B_12) or folic acid deficiency
  * Gastrointestinal bleeding within the past 2 weeks
  * Hemolysis
  * Myelodysplastic syndromes, myeloproliferative disorders, or acute myeloid leukemia
* No primary hematologic disorder causing chronic moderate to severe anemia (e.g., congenital dyserythropoietic anemia, homozygous hemoglobin S disease or compound heterozygous sickling states, or thalassemia major)

  * Carriers of these disease states allowed provided they are not anemic prior to cancer diagnosis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* Not pregnant or nursing

  * No delivery of a baby of ≥ 18 weeks estimated gestational age within the past 3 months (90 days)
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight > 40.0 kg and < 150.0 kg
* No known hypersensitivity to epoetin alfa, darbepoetin alfa, mammalian-cell derived products, or human albumin
* No uncontrolled hypertension, defined as systolic blood pressure (BP) ≥ 180 mm Hg and/or diastolic BP ≥ 100 mm Hg, despite medical therapy
* No pulmonary emboli and/or deep vein thrombosis within the past 12 months

  * Patients actively receiving warfarin for a minimum of 4 weeks are exempted from this requirement
  * Prior superficial thrombophlebitis allowed
* No cerebrovascular accident, ischemic stroke, acute coronary syndrome (e.g., unstable angina or Q-wave or non-Q wave myocardial infarction), or other arterial or venous thrombotic events within the past 6 months
* No history of chronic hypercoagulable disorders (e.g., activated protein C resistance, anti-cardiolipin disorder, protein C deficiency, or protein S deficiency)

  * Patients receiving anticoagulation therapy (warfarin or acetylsalicyclic acid [aspirin] at a dose of ≥ 325 mg/day) for these conditions are eligible provided therapy is continued during the study period
* History of previously treated seizures allowed provided the patient has been seizure-free for a minimum of 3 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 1 year since prior peripheral blood stem cell, bone marrow, or cord blood transplantation
* More than 14 days since prior red blood cell transfusion
* More than 14 days since prior major surgery, including, but not limited to, any of the following:

  * Amputation
  * Invasion of a body cavity or of the central nervous system using a scalpel, saw, or laser cutting tool
  * Resection of a body part (or parts), whether solid or liquid tissue or both, that includes ≥ 1% of a patient's preoperative weight
  * The following are not considered major surgery:

    * Diagnostic/therapeutic thoracentesis or paracentesis
    * Diagnostic skin biopsy
    * Digit or fingernail/thumbnail resection or laceration repair under local anesthesia
    * Diagnostic fat aspiration
    * Otic irrigation to remove cerumen impaction
    * Tympanocentesis
    * Uncomplicated dental extraction
    * Uncomplicated tonsillectomy
    * Laser corneal remodeling for refraction purposes
    * Cosmetic or therapeutic eyelid surgery
    * Bone marrow aspiration and biopsy
* More than 10 weeks since prior darbepoetin alfa, epoetin alfa, or any investigational form of erythropoietin (e.g., gene-activated erythropoietin or novel erythropoiesis stimulating protein)
* No planned stem cell transplantation within the next 4 months (18 weeks)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred and thirty-nine (239) participants were enrolled at 10 Mayo Clinic Cancer Research Consortium (MCCRC) sites between February 2007 and December 2008.
Pre-assignment Details: There were two canceled participants and 1 ineligible participants prior to study medication begins. These three participants were excluded from all analysis.
Groups:
- Epoetin Alfa - 40k Weekly: Patients receive Epoetin alfa 40,000 units subcutaneously every week for 15 weeks (15 doses)
- Epoetin Alfa - 80k Every 3 Weeks: Patients receive Epoetin alfa 80,000 units subcutaneously every 3 weeks for 15 weeks (5 doses)
- Epoetin Alfa - 120k Every 3 Weeks: Patients receive Epoetin alfa 120,000 units subcutaneously every 3 weeks for 15 weeks (5 doses)
- Darbepoetin Alfa - 500 mcg Every 3 Weeks: Patients receive Darbepoetin alfa 500 micrograms (mcg) subcutaneously every 3 weeks for 15 weeks (5 doses)
Period: Overall Study
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Started | 61 | 60 | 58 | 57
Completed | 39 | 33 | 40 | 40
Not Completed | 22 | 27 | 18 | 17
Not completed — Withdrawal by Subject | 1 | 6 | 4 | 9
Not completed — Death | 4 | 7 | 7 | 1
Not completed — Adverse Event | 8 | 3 | 2 | 2
Not completed — Other | 8 | 11 | 5 | 5
Not completed — Cancel | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were evaluable per protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks | Total
Number analyzed (Participants) | 61 | 60 | 58 | 57 | 236
Age, Continuous [Median (Full Range); unit: years] | 65.0 [44.0 to 94.0] | 68.0 [37.0 to 91.0] | 65.0 [19.0 to 81.0] | 67.0 [40.0 to 89.0] | 66.0 [19.0 to 94.0]
Gender [Count of Participants; unit: Participants]
  Female | 37 | 24 | 33 | 42 | 136
  Male | 24 | 36 | 25 | 15 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 5 | 14
  White | 58 | 57 | 52 | 52 | 219
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 58 | 57 | 236
Anemia [Number; unit: participants]
  Mild: Hemoglobin of 9.5-11 | 45 | 43 | 43 | 42 | 173
  Severe: Hemoglobin < 9.5 | 16 | 17 | 15 | 15 | 63
Platinum Containing Regimen [Number; unit: participants]
  Yes | 27 | 27 | 27 | 25 | 106
  No | 34 | 33 | 31 | 32 | 130
Primary Tumor Type [Number; unit: participants]
  Hematologic | 5 | 6 | 5 | 4 | 20
  Solid Tumor | 56 | 54 | 53 | 53 | 216
Height [Median (Full Range); unit: cm] | 167.6 [149.7 to 193.0] | 168.0 [154.0 to 201.0] | 165.2 [150.0 to 190.0] | 166.5 [152.4 to 187.0] | 167.0 [149.7 to 201.0]
Baseline Hemoglobin [Median (Full Range); unit: g/dL] | 10.1 [7.8 to 10.6] | 9.9 [8.4 to 10.5] | 9.9 [7.7 to 10.5] | 9.9 [7.4 to 10.5] | 9.9 [7.4 to 10.6]
Weight [Median (Full Range); unit: kg] | 69.1 [44.5 to 125.4] | 72.6 [51.3 to 133.0] | 70.6 [44.1 to 120.0] | 71.0 [42.5 to 141.0] | 71.3 [42.5 to 141.0]

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Who Exhibit a Hematopoietic Response
Description: A hematopoietic response was defined as Hb rise >2 g/dL from baseline or achieving Hb ≥ 11.5 g/dL, whichever occurs first, in the absence of RBC transfusions within 14 days of measurement) during the treatment period
Time Frame: 20 weeks
Population: All patients that were evaluable per protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
Percentage of participants | 68.9 | 61.7 | 65.5 | 66.7
Statistical Analysis 1: Comparison: Epoetin Alfa - 40k Weekly vs Epoetin Alfa - 80k Every 3 Weeks vs Epoetin Alfa - 120k Every 3 Weeks vs Darbepoetin Alfa - 500 mcg Every 3 Weeks; With 80 patients per treatment arm, there will be> about 80% power to detect a difference through Fisher's exact test across two> treatment arms of 25% in the true percentage of patients that experience a> hematopoietic response as defined previously, if that percentage is at least 30% in> the superior group, again with a 1.7% type I error rate; Test type: Non-Inferiority or Equivalence — If the hematopoietic response rate in the standard therapy group is far from 50% (<25% or >75%), the> above sample size will provide an 80% power to detect a difference as small as> 25%; p > 0.41, Fisher Exact

2. Secondary Outcome: Weekly Change in Hemoglobin Levels
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and an every-3-weeks darbepoetin alfa schedule
Time Frame: Baseline and Week 4, 7, 10, 13, 16
Population: All patients that were evaluable per protocol and had hemoglobin data at baseline, week 4, 7, 10, 13 or 16.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
g/dL
  Week 4 Minus Baseline | 1.0 (1.26) | 0.6 (1.02) | 0.7 (1.21) | 0.4 (1.21)
  Week 7 Minus Baseline | 1.7 (1.28) | 1.0 (1.58) | 1.1 (1.25) | 1.5 (1.59)
  Week 10 Minus Baseline | 1.7 (1.39) | 1.2 (1.42) | 1.2 (1.37) | 1.5 (1.44)
  Week 13 Minus Baseline | 2.1 (1.27) | 1.2 (1.51) | 1.3 (1.32) | 1.6 (1.65)
  Week 16 Minus Baseline | 1.7 (1.67) | 1.2 (1.64) | 1.6 (1.44) | 1.9 (1.41)

3. Secondary Outcome: Time Required to Achieve Hemoglobin Levels >= 11.5 g/dL
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule
Time Frame: 16 weeks
Population: All patients that were evaluable per protocol and had hemoglobin levels data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
days | 32 [28 to 37] | 50 [35 to 68] | 49 [35 to 77] | 49 [35 to 64]
Statistical Analysis 1: Comparison: Epoetin Alfa - 40k Weekly vs Epoetin Alfa - 80k Every 3 Weeks vs Epoetin Alfa - 120k Every 3 Weeks vs Darbepoetin Alfa - 500 mcg Every 3 Weeks; Test type: Non-Inferiority or Equivalence — A sample size of 80 patients per arm will provide> 80% power to detect differences between average hemoglobin levels in the> reference arm and another treatment of 50% of the standard deviation. Note that> typically one would expect the estimates for the standard deviation at a single time> point to differ from the standard deviation for the difference from baseline; p > 0.13, Fisher Exact

4. Secondary Outcome: Mean Hemoglobin Change From Week 1 to Week 16
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and an every-3-weeks darbepoetin alfa schedule. The positive numbers represent hemoglobin increases and negative numbers represent hemoglobin decreases.
Time Frame: Week 1 and Week 16
Population: All patients that were evaluable per protocol and had hemoglobin data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
g/dL | 11.0 (1.03) | 10.3 (1.04) | 10.6 (0.8) | 10.7 (0.96)

5. Secondary Outcome: The Percentage of Participants Requiring Red Blood Cell (RBC) Transfusions
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule
Time Frame: 16 weeks
Population: All patients that were evaluable per protocol and had RBC transfusions data.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
percentage of participants | 27.9 | 33.3 | 22.4 | 29.8
Statistical Analysis 1: Comparison: Epoetin Alfa - 40k Weekly vs Epoetin Alfa - 80k Every 3 Weeks vs Epoetin Alfa - 120k Every 3 Weeks vs Darbepoetin Alfa - 500 mcg Every 3 Weeks; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.49, Fisher Exact

6. Secondary Outcome: The Total RBC Transfusion Needed
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule
Time Frame: 16 weeks
Population: All patients that were evaluable per protocol and had RBC transfusions data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
g/dL | 1.1 (2.33) | 1.2 (2.67) | 0.6 (1.20) | 1.1 (2.31)

7. Secondary Outcome: The Percentage of Participants With Dose Omitted Due to Hematologic Reason
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule
Time Frame: 16 Weeks
Population: All patients that were evaluable per protocol.
Measure: Number; unit: percentage of Participants
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
percentage of Participants | 63.9 | 30 | 34.5 | 45.6

8. Secondary Outcome: The Percentage of Participants Reported Grade 3 or 4 Adverse Events
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule. Adverse events were measured by Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Time Frame: 16 weeks
Population: All patients that were evaluable per protocol and reported at least one value after baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 60 | 60 | 58 | 55
percentage of participants | 22 | 22 | 17 | 13
Statistical Analysis 1: Comparison: Epoetin Alfa - 40k Weekly vs Epoetin Alfa - 80k Every 3 Weeks vs Epoetin Alfa - 120k Every 3 Weeks vs Darbepoetin Alfa - 500 mcg Every 3 Weeks; With 80 patients per treatment arm, there will be about 80% power to detect a difference through Fisher's exact test across two treatment arms of 25% in the true percentage of patients that experience a hematopoietic response as defined previously, if that percentage is at least 30% in the superior group, again with a 1.7% type I error rate; Test type: Non-Inferiority or Equivalence — If the hematopoietic response rate in the standard therapy group is far from 50% (<25% or >75%), the above sample size will provide an 80% power to detect a difference as small as 25%; p > 0.56, Fisher Exact

9. Secondary Outcome: Quality of Life as Measured by Functional Assessment of Cancer Therapy Scales for Anemia (FACT-AN) Over All Follow-up Evaluations
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule. FACT-AN consist of Fatigue concerns subscale and non-fatigue concerns subscale. FACT Total Anemia score was calculated by adding the two subscales scores and transformed into 0-100 scale. FACT Total Anemia, Fatigue concerns scale and Non-Fatigue concerns scale are all ranges: 0 (Worst QOL) to 100 (Best QOL). Average scores across all time points for each subscale and total scale were calculated.
Time Frame: Weeks 4, 7, 10, 13 and 16
Population: All patients that were evaluable per protocol with QOL data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
units on a scale
  FACT Fatigue Concerns | 48.6 (17.13) | 52.0 (20.75) | 52.6 (23.12) | 49.8 (19.66)
  FACT Nonfatigue Concerns | 60.6 (13.08) | 62.2 (16.64) | 61.3 (16.27) | 59.4 (13.39)
  FACT Total Anemia | 52.8 (14.58) | 55.6 (18.08) | 55.6 (19.85) | 53.1 (16.24)

10. Secondary Outcome: Quality of Life as Measured by Linear Analogue Self Assessment Over All Follow-up Evaluation
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule. Linear Analogue Self Assessment (LASA) consists of 10 single-item numeric analogue scales on a scale of 0 to 10. Higher scores indicate better quality of life (QOL) on overall QOL, mental, physical, emotional spiritual QOL and Social activity; and constant pain, highest pain severity, level of fatigue and anxiety. Average scores across all time points for each item were calculated.
Time Frame: Weeks 4, 7, 10, 13 and 16
Population: All patients that were evaluable per protocol with QOL data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
units on a scale
  Overall QOL | 6.4 (1.59) | 6.5 (2.00) | 6.6 (2.17) | 6.1 (1.61)
  Mental QOL | 6.9 (1.80) | 7.0 (1.97) | 7.2 (1.91) | 6.5 (1.39)
  Physical QOL | 5.7 (1.54) | 5.8 (2.11) | 5.9 (2.22) | 5.8 (1.65)
  Emotional QOL | 6.5 (1.68) | 6.8 (1.99) | 6.7 (2.03) | 6.3 (1.80)
  Social Activity Level | 5.5 (2.08) | 5.5 (2.12) | 5.4 (2.34) | 5.1 (2.01)
  Spiritual QOL | 7.4 (1.54) | 7.4 (1.81) | 7.3 (2.07) | 6.8 (1.99)
  Pain Frequency | 4.5 (2.46) | 4.3 (2.96) | 3.9 (3.02) | 4.2 (2.42)
  Pain Severity | 4.1 (2.16) | 3.8 (2.72) | 3.7 (2.88) | 4.0 (2.24)
  Fatigue | 5.6 (1.59) | 5.5 (2.02) | 5.6 (2.14) | 5.4 (1.60)
  Anxiety | 4.1 (1.81) | 3.9 (2.20) | 4.6 (2.36) | 4.2 (1.67)

11. Secondary Outcome: Quality of Life as Measured by Brief Fatigue Inventory Overall All Follow-up Evaluations
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule. Brief Fatigue Inventory (BFI) consist of 3 single-item numeric analogue scales on a scale of 0 to 10; and an interference scale formed by 6 single-item numeric scales on a scale of 0 to 10. Higher scores indicate fatigue as bad as you can imagine for fatigue now, usual fatigue and worse fatigue; and completely interferes for BFI interference. Average scores across all time points for fatigue now, usual fatigue, worst fatigue and BFI interference subscale were calculated.
Time Frame: Weeks 4, 7, 10, 13 and 16
Population: All patients that were evaluable per protocol with QOL data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
units on a scale
  Fatigue Now | 4.8 (2.25) | 4.6 (2.44) | 4.6 (2.53) | 4.7 (2.25)
  Usual Fatigue | 4.7 (2.12) | 4.7 (2.40) | 4.7 (2.53) | 4.7 (2.24)
  Worst Fatigue | 5.5 (2.17) | 5.6 (2.54) | 5.4 (2.60) | 5.3 (2.43)
  BFI Interference | 4.3 (1.95) | 4.1 (2.42) | 4.3 (2.60) | 4.4 (2.17)

12. Secondary Outcome: Quality of Life as Measured by Symptom Distress Scale (SDS) Over All Follow-up Evaluations
Description: To compare the effects of the 3 different epoetin alfa dosing schedules and a darbepoetin alfa schedule. SDS Scale range: 1 (No Symptom), 5 (Worst Symptom). Average scores across all time points for each item were calculated.
Time Frame: Weeks 4, 7, 10, 13 and 16
Population: All patients that were evaluable per protocol with QOL data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Number analyzed (Participants) | 61 | 60 | 58 | 57
units on a scale
  Nausea Frequency | 1.6 (0.64) | 1.5 (0.67) | 1.6 (0.56) | 1.6 (0.73)
  Nausea Severity | 1.5 (0.59) | 1.4 (0.62) | 1.4 (0.61) | 1.6 (0.73)
  Appetite | 2.3 (0.96) | 2.3 (0.94) | 2.2 (0.98) | 2.4 (0.91)
  Insomnia | 2.4 (0.99) | 2.0 (0.88) | 2.3 (0.89) | 2.4 (0.91)
  Pain Frequency | 2.7 (1.12) | 2.5 (1.15) | 2.4 (1.22) | 2.7 (1.16)
  Pain Severity | 2.2 (0.97) | 2.0 (1.02) | 2.0 (1.05) | 2.1 (0.88)
  Fatigue | 3.1 (0.82) | 3.0 (0.94) | 2.8 (0.97) | 2.9 (0.91)
  Bowel | 2.2 (1.00) | 2.4 (1.20) | 2.3 (1.05) | 2.3 (0.95)
  Concentration | 2.2 (0.99) | 2.0 (1.00) | 1.9 (0.89) | 2.2 (0.96)
  Appearance | 2.1 (0.89) | 2.2 (1.05) | 2.0 (1.09) | 2.2 (0.97)
  Breathing | 1.5 (0.54) | 1.6 (0.64) | 1.6 (0.82) | 1.7 (1.01)
  Outlook | 2.2 (0.98) | 2.1 (0.99) | 2.1 (0.91) | 2.4 (1.02)
  Cough | 1.8 (0.77) | 1.7 (0.66) | 1.8 (0.69) | 2.0 (0.84)
  Depression | 1.8 (0.64) | 1.7 (0.79) | 1.8 (0.65) | 2.0 (0.90)

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: All evaluable patients per protocol that reported at least one value after baseline.
Arm/Group | Epoetin Alfa - 40k Weekly | Epoetin Alfa - 80k Every 3 Weeks | Epoetin Alfa - 120k Every 3 Weeks | Darbepoetin Alfa - 500 mcg Every 3 Weeks
Serious Adverse Events (participants affected / at risk) | 4/60 | 7/60 | 4/58 | 2/56
Other Adverse Events (participants affected / at risk) | 21/60 | 16/60 | 16/58 | 7/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoetin Alfa - 40k Weekly (N=60) | Epoetin Alfa - 80k Every 3 Weeks (N=60) | Epoetin Alfa - 120k Every 3 Weeks (N=58) | Darbepoetin Alfa - 500 mcg Every 3 Weeks (N=56)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epoetin Alfa - 40k Weekly (N=60) | Epoetin Alfa - 80k Every 3 Weeks (N=60) | Epoetin Alfa - 120k Every 3 Weeks (N=58) | Darbepoetin Alfa - 500 mcg Every 3 Weeks (N=56)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 5 (6) | 3 (3) | 2 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Fatigue (General disorders) | 3 (3) | 4 (12) | 4 (6) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (5) | 2 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal pelvis fistula (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes